CLINICAL TRIAL: NCT00005982
Title: Phase II Study of 506U78 (NSC #686673) in Patients With Previously Treated Cutaneous T-Cell Lymphoma
Brief Title: 506U78 in Treating Patients With Recurrent or Refractory Cutaneous T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02344; ID99-213; CDR0000067970 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — nelarabine

ARMS (1):
- Treatment (nelarabine) (Experimental): Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment continues every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: nelarabine; Other: pharmacological study

INTERVENTIONS:
Drug: nelarabine — Given IV
  Other Names: 506U78; Arranon; GW506U78
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Phase II trial to study the effectiveness of 506U78 in treating patients who have recurrent or refractory cutaneous T-cell lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, failure-free survival, and progression-free survival of patients with recurrent or refractory cutaneous T-cell lymphoma treated with 506U78.

II. Determine the toxicity of this drug in these patients. III. Study the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment continues every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory cutaneous T-cell lymphoma

  * Large cell transformation of cutaneous T-cell lymphoma allowed
* No active CNS disease
* Performance status - Zubrod 0-2
* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 100,000/mm^3*
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGPT no greater than 2.5 times ULN
* Creatinine clearance greater than 50 mL/min
* No history of symptomatic cardiac dysfunction
* No history of pericardial effusion
* HIV negative
* No grade 2 or greater sensory or motor neuropathy
* No history of seizures
* No other malignancy within the past 5 years except curatively treated basal cell carcinoma of the skin of carcinoma in situ of the cervix
* No medical, psychiatric, or social condition that would preclude study
* No other concurrent serious illness or active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior stem cell or bone marrow transplantation (BMT)
* No more than 1 prior immunotherapy regimen
* No more than 3 prior systemic regimens with denileukin diftitox
* At least 3 weeks since prior biologic therapy
* No concurrent BMT
* No prior 506U78
* No more than 3 prior systemic chemotherapy regimens comprising any of the following:

  * Oral methotrexate
  * Topical mechlorethamine
* At least 3 weeks since prior chemotherapy
* No other concurrent chemotherapy
* At least 3 weeks since prior anticancer endocrine therapy
* No concurrent topical or systemic steroids
* At least 3 weeks since prior radiotherapy
* No more than 3 prior systemic regimens comprising any of the following:

  * Total skin electron beam therapy
  * Spot radiotherapy
* No more than 3 prior systemic regimens comprising any of the following:

  * Oral retinoids
  * Ultraviolet therapy (PUVA)
* At least 3 weeks since prior anticancer therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-04; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) defined as CR + PR rates | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States